CLINICAL TRIAL: NCT00200902
Title: Factors of Treatment Response in Major Depressive Disorder
Brief Title: Evaluation of Depression Symptoms and Brain Activity Associated With Response to Treatment of Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Eli Lilly and Company (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AT002479-02 (NIH); R01AT002479-02 (NIH); 04-02-068
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Depression
Keywords: Major depressive disorder; MDD; Antidepressant
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride; Duloxetine Hydrochloride; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MED (Active Comparator): For medication treatment, three different types were utilized and assigned specifically to each subject depending on their condition:
  MED 1: Venlafaxine XR. MED 2: Duloxetine (Cymbalta) MED 3: Escitalopram (Lexapro)
  Interventions: Drug: Venlafaxine (Effexor), Duloxetine (Cymbalta), Escitalopram (Lexapro)
- Placebo (PBO) (Placebo Comparator): Subjects enrolled will receive interpersonal clinical interaction (ICI) along with a placebo treatment (Interaction and assessment as in ICI plus double blinded treatment with placebo tablets).
  Interventions: Other: Placebo
- Interpersonal Clinical Interaction (ICI) (Other): Subjects assigned to the interpersonal clinical interaction (ICI) will undergo a one-week waiting period after the initial assessment. Visits will involve a session with a research nurse that will be approximately 20 minutes in length; visits at baseline, end of lead-in, and 1, 2, 4, and 8 weeks also will include a brief (5-10 minutes) meeting with a physician.
  Interventions: Behavioral: Interpersonal Clinical Interaction (ICI)

INTERVENTIONS:
Drug: Venlafaxine (Effexor), Duloxetine (Cymbalta), Escitalopram (Lexapro) — Subjects assigned to the placebo (PBO) or medication (MED) condition will enter double-blind treatment with either venlafaxine XR, duloxetine, escitalopram, or placebo after lead-in. They will undergo the same schedule, structure, and intensity of visits as in the ICI condition, but also will be randomized to receive treatment with a pill. Subjects randomized to medication will be started on one tablet each morning of either venlafaxine XR 75 mg., duloxetine 30 mg., or escitalopram 10 mg. Dosages will be increased in a double-blinded manner by increasing the number of pills administered by one pill every three to five days until the final dose is achieved (225 mg., 90 mg., and 30 mg. respectively for venlafaxine XR, duloxetine, and escitalopram). In order to maintain blinding during dosage increase, the number of tablets of placebo will be increased every three to five days as well.
  Arms: MED
Other: Placebo — Subjects assigned to the placebo (PBO) or medication (MED) condition will enter double-blind treatment with either venlafaxine XR, duloxetine, escitalopram, or placebo after lead-in. They will undergo the same schedule, structure, and intensity of visits as in the ICI condition, but also will be randomized to receive treatment with a pill. Subjects randomized to medication will be started on one tablet each morning of either venlafaxine XR 75 mg., duloxetine 30 mg., or escitalopram 10 mg. Dosages will be increased in a double-blinded manner by increasing the number of pills administered by one pill every three to five days until the final dose is achieved (225 mg., 90 mg., and 30 mg. respectively for venlafaxine XR, duloxetine, and escitalopram). In order to maintain blinding during dosage increase, the number of tablets of placebo will be increased every three to five days as well.
  Arms: Placebo (PBO)
Behavioral: Interpersonal Clinical Interaction (ICI) — Interaction with and assessment by clinical research personnel on a fixed schedule, with the pharmacotherapeutic alliance assessed both by research personnel and subjects.
  Arms: Interpersonal Clinical Interaction (ICI)

SUMMARY:
This study will use measurements of depression symptoms and brain activity to determine what factors may influence an individual's response to treatment for depression.

DETAILED DESCRIPTION:
We are using depression symptom measurements and measurements of brain electrical activity (EEG) to determine what factors may influence whether a patient is likely to show a response to antidepressant medication, placebo, or only clinical visits (without the use of pills) during a treatment trial for depression.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unipolar major depression

Exclusion Criteria:

* Substance abuse
* Psychotic disorder
* History of severe head trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F. Leuchter, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Laboratory of Brain, Behavior, and Pharmacology, Los Angeles, California, United States

REFERENCES:
- [Derived] Leuchter AF, Hunter AM, Tartter M, Cook IA. Role of pill-taking, expectation and therapeutic alliance in the placebo response in clinical trials for major depression. Br J Psychiatry. 2014 Dec;205(6):443-9. doi: 10.1192/bjp.bp.113.140343. Epub 2014 Sep 11. PMID 25213159
- See also: Depression Research - Click here for more information about this study: Psychobiologic Factors of the Placebo Response in MDD — http://www.DepressionResearch.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 133 subjects were screened for eligibility and 88 were eligible for enrollment between 8/19/05 - 8/7/08 at the UCLA Laboratory of Brain, Behavior, and Pharmacology. 88 participants were randomized however, n=67 for many of the measures as subjects who did not complete the Week 8 visit were not included in the analysis.
Pre-assignment Details: Subjects were required to wash out of any other antidepressant medications for one week (30 days if washing out from fluoxetine).
Groups:
- MEDS + ICI: MED 1-venlafaxine XR, MED 2-Duloxetine (Cymbalta), MED 3-Escitalopram (Lexapro)
- ICI Alone: Subjects assigned to the interpersonal clinical interaction (ICI). Visits will involve a session with a research nurse that will be approximately 20 minutes in length; visits at baseline, end of lead-in, and 1, 2, 4, and 8 weeks also will include a brief (5-10 minutes) meeting with a physician.
Period: Overall Study
Arm/Group | MEDS + ICI | Placebo+ICI | ICI Alone
Started (Overall for this study, n=67 assessed for many measures in Results section.) | 39 | 29 | 20
Completed | 29 | 26 | 12
Not Completed | 10 | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Medication Treatment (MED): MED 1-venlafaxine XR, MED 2-Duloxetine (Cymbalta), MED 3-Escitalopram (Lexapro)
- Interpersonal Clinical Interaction: Subjects assigned to the interpersonal clinical interaction (ICI). Visits involve a session with a research nurse that will be approximately 20 minutes in length; visits at baseline, end of lead-in, and 1, 2, 4, and 8 weeks also will include a brief (5-10 minutes) meeting with a physician.
- Total: Total of all reporting groups
Arm/Group | Medication Treatment (MED) | Placebo | Interpersonal Clinical Interaction | Total
Number analyzed (Participants) | 39 | 29 | 20 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 29 | 20 | 88
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.67 (13.63) | 41.75 (14.35) | 43.1 (12.7) | 41.96 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 12 | 55
  Male | 14 | 11 | 8 | 33
Region of Enrollment [Number; unit: participants]
  United States | 29 | 26 | 12 | 67

OUTCOME MEASURES:

1. Primary Outcome: Response as Assessed by Participants' Change in Depression Rating
Description: Comparison of treatment arms (Medication + ICI, Placebo+ICI, and ICI only). The Hamilton Depression Rating Scale (HAM-D-17) used here is a 17-item scale that measures severity of depression. Items are individually scored from 0-4 or from 0-2 depending on the item, and the individual scores for each item are added to comprise one score. Higher scores indicate greater severity of depression. Possible scores on the scale range from a minimum of zero (0) to a maximum of 52.Response is defined as a 50% decrease in HAMD-17 scoring. Remission defined as a HAMD-17 score of 7 or less.
Time Frame: Baseline, Week 8
Population: Participants completing the Week 8 visit were included in the analysis (n=67)
Measure: Count of Participants; unit: Participants
Groups:
- MEDICATIONS: Three different types of medications were utilized and assigned specifically to each subject depending on their condition. Interpersonal clinical interaction (ICI) plus clinically assigned medication (Venlafaxine XR, Duloxetine, or Escitalopram).
- Placebo (PBO): Interpersonal clinical interaction (ICI) plus placebo
- Interpersonal Clinical Interaction (ICI): Interpersonal clinical interaction (ICI) ONLY
Arm/Group | MEDICATIONS | Placebo (PBO) | Interpersonal Clinical Interaction (ICI)
Number analyzed (Participants) | 29 | 26 | 12
Participants
  Responders | 17 | 11 | 1
  Remitters | 9 | 9 | 0

2. Primary Outcome: Average Change in 3 Weeks of Participant Treatment Expectations
Description: Patient Attitudes and Expectations Form used for assessing expectation. The California Pharmacotherapy Alliance Scale, a measure associated with outcomes of antidepressant pharmacotherapy, used to measure participants' perceptions of: (a) participants' commitment to treatment; (b) participants' working capacity; (c) treatment providers' understanding and involvement; and (d) goal and working strategy consensus between participant and treatment provider. This is a 24-item questionnaire with a 7-point Likert scale (1 = not at all, 7 = very much so). Total score ranges from a minimum of 0 and a maximum of 120. The score is determined by a combination of negative and positive items. To assure negative items are reflected, subtract each of the negative item ratings from 8; for example, a rating of 1 becomes 7 (8 minus 1). The scores are computed by summing the items and dividing the total by 6 to procure the mean rating. A lower score indicates a worse outcome.
Time Frame: Averaged over 3 time points (Baseline, randomization, and end of lead-in)
Population: 88 participants who completed the first 3 time points in the study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Medication (MED): MED 1-venlafaxine XR, MED 2-Duloxetine (Cymbalta), MED 3-Escitalopram (Lexapro)
- Placebo (PBO): Placebo subjects received interpersonal clinical interaction (ICI) along with placebo treatment.
  Placebo: Subjects assigned to the placebo (PBO) or medication (MED) condition entered double-blind treatment with either venlafaxine XR, duloxetine, escitalopram, or placebo after lead-in. They underwent the same schedule, structure, and intensity of visits as in the ICI condition, but also were randomized to receive treatment with a pill. Subjects randomized to medication started on one tablet each morning of either venlafaxine XR 75 mg., duloxetine 30 mg., or escitalopram 10 mg. Dosages will be increased in a double-blinded manner by increasing the number of pills administered by one pill every three to five days until the final dose is achieved (225 mg., 90 mg., and 30 mg. respectively for venlafaxine XR, duloxetine, and escitalopram). In order to maintain blinding during dosage increase, the number of tablets of placebo will be increased every three to five days as well.
Arm/Group | Medication (MED) | Placebo (PBO) | Interpersonal Clinical Interaction (ICI)
Number analyzed (Participants) | 39 | 29 | 20
units on a scale | 3.55 (.78) | 3.94 (.61) | 3.17 (1.16)

3. Primary Outcome: Change in Hamilton Depression Assessment Score
Description: Comparison of treatment arms (Medication + ICI, Placebo+ICI, and ICI only). The Hamilton Depression Rating Scale used here is a 17-item scale that measures severity of depression. Items are individually scored from 0-4 or from 0-2 depending on the item, and the individual scores for each item are added to comprise one score. Higher scores indicate greater severity of depression/worse outcome. Possible scores on the scale range from a minimum of zero (0) to a maximum of 52.
Time Frame: Baseline,Week 8
Measure: Mean (Standard Deviation); unit: HAMD score
Groups:
- Medication (MED): Venlafaxine (Effexor), Duloxetine (Cymbalta), or Escitalopram (Lexapro) + ICI
- Placebo (PBO): Placebo + ICI
- Interpersonal Clinical Interaction (ICI): ICI ONLY
Arm/Group | Medication (MED) | Placebo (PBO) | Interpersonal Clinical Interaction (ICI)
Number analyzed (Participants) | 29 | 26 | 12
HAMD score
  Percent Change in HAM-D | -0.46 (0.31) | -0.36 (0.39) | -0.05 (0.27)
  Change in HAM-D | -10.05 (6.60) | -7.59 (7.98) | -1.37 (5.27)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Medication: Venlafaxine (Effexor), Duloxetine (Cymbalta), or Escitalopram (Lexapro) + ICI
Arm/Group | Medication | Placebo (PBO) | Interpersonal Clinical Interaction (ICI)
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/29 | 0/20
Other Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/12

LIMITATIONS AND CAVEATS:
Individuals entering this study were aware that they might be assigned to a treatment condition that did not involve the use of medication; it is not certain that they are representative of people with MDD who would enter clinical trials for MDD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No